CLINICAL TRIAL: NCT01601535
Title: Phase I/II Study of MLN8237 in Combination With Irinotecan and Temozolomide for Patients With Relapsed or Refractory Neuroblastoma
Brief Title: Study of MLN8237 in Combination With Irinotecan and Temozolomide
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New Approaches to Neuroblastoma Therapy Consortium (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: N2009-03
Record Dates: First submitted 2012-05-11; First posted 2012-05-18 (Estimated); Results first posted 2019-07-31 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — MLN 8237; Irinotecan; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Every course will be 21 days. MLN8237 will be administered orally daily starting on day 1 through day 7.
  Irinotecan will be administered intravenously during each course on study day 1 through day 5.
  Temozolomide will be administered orally during each course on study day 1 through day 5.
  Interventions: Drug: MLN8237; Drug: Irinotecan; Drug: Temozolomide

INTERVENTIONS:
Drug: MLN8237 — Every course will be 21 days. MLN8237 will be administered orally daily starting on day 1 through day 7.
Drug: Irinotecan — Irinotecan will be administered intravenously during each course on study day 1 through day 5.
  Other Names: Camptosar
Drug: Temozolomide — Temozolomide will be administered orally during each course on study day 1 through day 5.
  Other Names: Temodar

SUMMARY:
The goal of the first part of this clinical trial (Phase I portion) is to study the side effects, drug breakdown (pharmacokinetics), and dosing of the drug MLN8237 when added to standard chemotherapy drugs, irinotecan and temozolomide.

The goal of the second part of this clinical trial (Phase II portion) is to learn how many children and young adults show improvements in their neuroblastoma when treated with the combination of MLN8237, irinotecan, and temozolomide.

DETAILED DESCRIPTION:
The Aurora A kinase has been shown to play an important role in neuroblastoma growth. Inhibition of Aurora A kinase activity attenuates the growth of neuroblastoma cells. MLN8237 is a selective small molecule inhibitor of Aurora A kinase that has completed pediatric single-agent phase I testing, as well as stage 1 phase 2 testing in patients with Neuroblastoma. MLN8237 showed activity against the NCI-sponsored Pediatric Preclinical Testing Program neuroblastoma in vivo panel that exceeded the activity level observed with chemotherapy agents routinely used in the treatment of neuroblastoma. Additional in vitro and in vivo studies have shown that Aurora A kinase inhibitors result in enhanced cytotoxicity when used in combination with chemotherapy. Irinotecan and temozolomide is a commonly used salvage regimen for patients with relapsed or refractory neuroblastoma. This combination has a modest objective response rate (16%) and is well-tolerated, suggesting that it will provide a useful platform for the study of novel compounds in combination with chemotherapy. Preclinical studies demonstrate marked enhancement of anti-neuroblastoma activity with the addition of MLN8237 to irinotecan and temozolomide. This study therefore evaluates the tolerability and activity of MLN8237 in combination with irinotecan and temozolomide in children with refractory or relapsed neuroblastoma. Patients receive irinotecan (50 mg/m2/dose IV) and temozolomide (100 mg/m2/dose orally) once daily for 5 days along with MLN8237 orally once daily for 7 days. The doses of irinotecan and temozolomide will be fixed and the dose of MLN8237 will be dose-escalated. In the phase I portion of the study, the primary aims are to determine the recommended phase II doses of this combination, describe the toxicity of this combination, and characterize the pharmacokinetic profile of MLN8237 and irinotecan when used in combination. In the phase II portion of the study, the primary aim is to determine the objective response rate of this combination in patients with relapsed or refractory neuroblastoma. With Amendment 5, the tolerability and pharmacokinetics of an MLN8237 oral solution will be evaluated. Optional correlative studies will evaluate UGT1A1 polymorphisms as predictors of toxicity and archival tumor tissue Aurora A expression as a predictor of response with this combination.

ELIGIBILITY:
Criteria that need to be met to participate in this study:

* Patients must be > 12 months and < 30 years of age when registered on study.
* Patients must have relapsed neuroblastoma, refractory neuroblastoma that had less than a partial response to standard treatment or persistent neuroblastoma that had at least a partial response to standard treatment. All patients must have at least ONE site of evaluable disease.

  o Patients who have at least a partial response to standard treatment who still have neuroblastoma that can be seen on CT/MRI or MIBG scans must have a surgical biopsy done of the tumor to confirm that it is neuroblastoma. Patients with relapsed or refractory neuroblastoma do not need to have a biopsy done to enter on study.
* Patients must have adequate heart, kidney, liver and bone marrow function. Patients who have bone marrow disease must still have adequate bone marrow function to enter the study.
* MLN8237 must be swallowed as whole tablets. Therefore, patients must be able to swallow pills to be eligible for study. One tablet is the size of small breath mint, or baby aspirin. Due to the size of MLN8237 tablets, patients must have a body surface area of at least 0.38 m2 to be eligible for study. A body surface area is a combination of a patient's height and weight. An example of a child with a BSA of 0.45 is a child that is 25 inches tall and weighs 25 pounds.You can use the link below to calculate your child's body surface area and determine if they are too small for this trial.

Patients cannot participate in the study if:

* Patients who have received prior MLN8237 are excluded from all phases of the study. Patients previously treated with irinotecan and/or temozolomide will be eligible if they have not had documented progressive disease during treatment with a regimen containing these agents.
* They have other medical problems that could get much worse if they had this treatment.
* They are on dialysis for bad kidney function.
* They are pregnant or breast feeding.
* They have active infections such as hepatitis or fungal infections.
* They have an allergy to treatment with cefixime and cefpodixime.
* They have brain metastasis at study entry, or have received cranial spinal radiation.
* They have had an allogeneic stem cell transplant (received stem cell from someone else).
* They can't cooperate with the special precautions that are needed for this trial.

Ages: 12 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2012-05; Primary Completion 2018-07-25 (Actual); Study Completion 2018-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven DuBois, MD, Study Chair — Dana-Farber Cancer Institute
Locations (13):
- United States (12):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Children Hospital of Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - University of Chicago Comer Children's Hospital, Chicago, Illinois
  - Childrens Hospital Boston, Dana-Farber Cancer Institute., Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
- Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] DuBois SG, Mosse YP, Fox E, Kudgus RA, Reid JM, McGovern R, Groshen S, Bagatell R, Maris JM, Twist CJ, Goldsmith K, Granger MM, Weiss B, Park JR, Macy ME, Cohn SL, Yanik G, Wagner LM, Hawkins R, Courtier J, Lai H, Goodarzian F, Shimada H, Boucher N, Czarnecki S, Luo C, Tsao-Wei D, Matthay KK, Marachelian A. Phase II Trial of Alisertib in Combination with Irinotecan and Temozolomide for Patients with Relapsed or Refractory Neuroblastoma. Clin Cancer Res. 2018 Dec 15;24(24):6142-6149. doi: 10.1158/1078-0432.CCR-18-1381. Epub 2018 Aug 9. PMID 30093449

RESULTS

PARTICIPANT FLOW:
Groups:
- DL 1: alisertib tablets (45 mg/m^2/dose x 7 days), irinotecan (50 mg/m^2/dose IV x 5 days), temozolomide (100 mg/m^2/dose orally x 5 days), myeloid growth factor support and cephalosporin diarrhea prophylaxis optional
- DL 1B: alisertib tablets (45 mg/m^2/dose x 7 days), irinotecan (50 mg/m^2/dose IV x 5 days), temozolomide (100 mg/m^2/dose orally x 5 days), myeloid growth factor support and cephalosporin diarrhea prophylaxis required
- DL 2B; Ph 2: alisertib tablets (60 mg/m^2/dose x 7 days), irinotecan (50 mg/m^2/dose IV x 5 days), temozolomide (100 mg/m^2/dose orally x 5 days), myeloid growth factor support and cephalosporin diarrhea prophylaxis required
- DL 3B: alisertib tablets (80 mg/m^2/dose x 7 days), irinotecan (50 mg/m^2/dose IV x 5 days), temozolomide (100 mg/m^2/dose orally x 5 days), myeloid growth factor support and cephalosporin diarrhea prophylaxis required
- Oral Solution: alisertib oral solution (45 mg/m^2/dose x 7 days), irinotecan (50 mg/m^2/dose IV x 5 days), temozolomide (100 mg/m^2/dose orally x 5 days), myeloid growth factor support and cephalosporin diarrhea prophylaxis required
Period: Phase 1
Arm/Group | DL 1 | DL 1B | DL 2B | DL 3B | Ph 2 | Oral Solution
Started | 6 | 6 | 6 | 4 | 0 | 0
Completed | 0 | 0 | 1 | 0 | 0 | 0
Not Completed | 6 | 6 | 5 | 4 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 2 | 0 | 0
Not completed — Progressive Disease | 2 | 3 | 2 | 1 | 0 | 0
Not completed — Started Another Treatment | 1 | 2 | 0 | 0 | 0 | 0
Period: Phase 2
Arm/Group | DL 1 | DL 1B | DL 2B | DL 3B | Ph 2 | Oral Solution
Started | 0 | 0 | 0 | 0 | 20 | 12
Completed | 0 | 0 | 0 | 0 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 19 | 12
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 5 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 8 | 2
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 5 | 7
Not completed — Started Another Treatment | 0 | 0 | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DL 1 | DL 1B | DL 2B | DL 3B | Ph 2 | Oral Solution | Total
Number analyzed (Participants) | 6 | 6 | 6 | 4 | 20 | 12 | 54
Age, Continuous [Median (Full Range); unit: years] | 8.60 [7.39 to 18.53] | 6.81 [4.70 to 13.26] | 7.67 [4.34 to 22.74] | 6.14 [4.66 to 12.66] | 10.74 [4.36 to 19.42] | 3.05 [1.69 to 7.20] | 7.61 [1.69 to 22.74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 1 | 6 | 6 | 16
  Male | 6 | 4 | 5 | 3 | 14 | 6 | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 0 | 1 | 0 | 0 | 1 | 0 | 2
  Not Hispanic Black or African American | 1 | 0 | 1 | 0 | 3 | 0 | 5
  Not Hispanic White | 5 | 5 | 5 | 4 | 14 | 12 | 45
  Not Hispanic Other | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Not Hispanic Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 4 | 20 | 12 | 54
Prior Irinotecan [Count of Participants; unit: Participants]
  Yes | 3 | 1 | 0 | 1 | 11 | 2 | 18
  No | 3 | 5 | 6 | 3 | 9 | 10 | 36
Prior Temozolomide [Count of Participants; unit: Participants]
  Yes | 3 | 1 | 0 | 1 | 10 | 2 | 17
  No | 3 | 5 | 6 | 3 | 10 | 10 | 37

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) When Given Together With Fixed Doses of Irinotecan and Temozolomide in Children and Young Adults With Relapsed or Refractory Neuroblastoma
Description: The MTD was the highest dose level tested at which fewer than two of six patients had first course DLT. Hematologic DLT was defined as grade 4 neutropenia for more than 7 days, need for platelet transfusion for a platelet count of less than 20,000/mL twice within a 7-day period, or greater than 14-day delay in the start of a subsequent course because of neutropenia or thrombocytopenia. Nonhematologic DLT was defined as any nonhematologic toxicity that delayed the start of a subsequent cycle by more than 14 days or any grade ≥3 toxicity with the exception of the following grade 3 toxicities: nausea, vomiting, anorexia, or dehydration resolving to grade ≤ 2 within 72 hours; increase in hepatic transaminase or electrolyte abnormality resolving to grade ≤ 1 within 7 days; diarrhea persisting for less than 72 hours; fever; infection; or febrile neutropenia. DLT definitions included only toxicities deemed at least possibly related to therapy.
Time Frame: 21 days, from study day 1
Measure: Number; unit: mg/m^2
Groups:
- Phase I: Patients received alisertib tablets at dose levels of 45, 60, and 80 mg/m^2 per day on days 1 to 7 along with irinotecan 50 mg/m^2 intravenously and temozolomide 100 mg/m^2 orally on days 1 to 5.
Arm/Group | Phase I
Number analyzed (Participants) | 22
mg/m^2 | 60

2. Primary Outcome: Dose Limiting Toxicity (DLT) Data Associated With the Determination of the Recommended Phase 2 Dose
Description: as for outcome 1
Time Frame: 21 days, from study day 1
Measure: Number; unit: DLTs
Arm/Group | DL 1 | DL 1B | DL 2B | DL 3B
Number analyzed (Participants) | 6 | 6 | 6 | 4
DLTs | 2 | 0 | 1 | 2

3. Primary Outcome: Pharmacokinetics When Given Together With Fixed Doses of Irinotecan and Temozolomide in Children and Young Adults With Relapsed or Refractory Neuroblastoma: Alisertib Day 4 Trough, Day 5 Trough and Cmax
Description: Outcomes included Alisertib, irinotecan, APC, SN-38, and SN-38G. APC, SN-38, and SN-38G are metabolites of irinotecan.
Time Frame: 1st week of cycle 1
Measure: Median (Full Range); unit: µM
Arm/Group | DL 1 | DL 1B | DL 2B | DL 3B | Oral Solution
Number analyzed (Participants) | 6 | 6 | 6 | 4 | 12
µM
  Alisertib Day 4 trough | 0.48 [0.09 to 0.98] | 0.35 [0.13 to 1.38] | 0.3 [0.22 to 4.07] | 0.73 [0.15 to 1.35] | 0.47 [0.09 to 3.37]
  Alisertib Day 5 trough | 0.37 [0.12 to 1.36] | 0.36 [0.18 to 0.65] | 0.2 [0.05 to 3.31] | 0.69 [0.25 to 1.27] | 0.58 [0.09 to 3.2]
  Alisertib Cmax | 2.56 [1.91 to 5.92] | 2.39 [1.72 to 5.92] | 3.77 [2.16 to 6.76] | 4.94 [3.99 to 6.22] | 8.66 [3.49 to 11.39]

4. Primary Outcome: Pharmacokinetics When Given Together With Fixed Doses of Irinotecan and Temozolomide in Children and Young Adults With Relapsed or Refractory Neuroblastoma: Alisertib Tmax and Half-life
Description: Outcomes included Alisertib, irinotecan, APC, SN-38, and SN-38G. APC, SN-38, and SN-38G are metabolites of irinotecan.
Time Frame: 1st week of cycle 1
Measure: Median (Full Range); unit: hour
Arm/Group | DL 1 | DL 1B | DL 2B | DL 3B | Oral Solution
Number analyzed (Participants) | 6 | 6 | 6 | 4 | 12
hour
  Alisertib Tmax | 2.04 [1.12 to 6.93] | 1.74 [0.65 to 2.9] | 2.5 [0.97 to 4] | 2.52 [2 to 3.03] | 2 [0.5 to 4]
  Alisertib Half-life | 7.20 [5.22 to 9.83] | 8.61 [4.2 to 18.2] | 6.19 [3.65 to 20.28] | 8.54 [5.35 to 10.05] | 8.34 [4.28 to 16.89]

5. Primary Outcome: Pharmacokinetics When Given Together With Fixed Doses of Irinotecan and Temozolomide in Children and Young Adults With Relapsed or Refractory Neuroblastoma: Alisertib AUC
Description: Outcomes included Alisertib, irinotecan, APC, SN-38, and SN-38G. APC, SN-38, and SN-38G are metabolites of irinotecan.
Time Frame: 1st week of cycle 1
Measure: Median (Full Range); unit: µM•hour
Arm/Group | DL 1 | DL 1B | DL 2B | DL 3B | Oral Solution
Number analyzed (Participants) | 6 | 6 | 6 | 4 | 12
µM•hour | 28.15 [16.9 to 65.5] | 21 [15.4 to 44.9] | 30.71 [19.61 to 117.03] | 47.73 [32.71 to 84.67] | 58.15 [32.03 to 144.72]

6. Primary Outcome: Pharmacokinetics When Given Together With Fixed Doses of Irinotecan and Temozolomide in Children and Young Adults With Relapsed or Refractory Neuroblastoma: Irinotecan Cmax, APC Cmax, SN-38 Cmax, and SN-38G Cmax
Description: Outcomes included Alisertib, irinotecan, APC, SN-38, and SN-38G. APC, SN-38, and SN-38G are metabolites of irinotecan.
Time Frame: 1st week of cycle 1
Measure: Median (Full Range); unit: ng/mL
Arm/Group | DL 1 | DL 1B | DL 2B | DL 3B | Ph 2 | Oral Solution
Number analyzed (Participants) | 6 | 6 | 6 | 4 | 12 | 8
ng/mL
  Irinotecan Cmax | 722 [502 to 880] | 703 [642 to 5,371] | 1,238 [493 to 1,757] | 784 [546 to 987] | 881 [490 to 1,757] | 732 [422 to 861]
  APC Cmax | 61.2 [23.1 to 480.4] | 59.8 [28.2 to 105] | 55.8 [25.7 to 76.3] | 43.4 [29.1 to 49.4] | 57.1 [25.7 to 132] | 51.4 [15.0 to 98.2]
  SN-38 Cmax | 9.5 [6.6 to 18.7] | 12.6 [5.8 to 16.5] | 12.0 [8.8 to 14.7] | 11.7 [7.0 to 13.8] | 10.4 [5.19 to 32.6] | 8.26 [4.62 to 33.1]
  SN-38G Cmax | 18.2 [16.0 to 46.9] | 16.9 [4.8 to 23.7] | 13.8 [7.0 to 26.8] | 13.0 [10.4 to 24.0] | 12.8 [6.96 to 50.5] | 15.2 [4.83 to 46.7]

7. Primary Outcome: Pharmacokinetics When Given Together With Fixed Doses of Irinotecan and Temozolomide in Children and Young Adults With Relapsed or Refractory Neuroblastoma: Irinotecan AUC, APC AUC, SN-38 AUC, and SN-38G AUC
Description: Outcomes included Alisertib, irinotecan, APC, SN-38, and SN-38G. APC, SN-38, and SN-38G are metabolites of irinotecan.
Time Frame: 1st week of cycle 1
Measure: Median (Full Range); unit: h·ng/mL
Arm/Group | DL 1 | DL 1B | DL 2B | DL 3B | Ph 2 | Oral Solution
Number analyzed (Participants) | 6 | 6 | 6 | 4 | 12 | 8
h·ng/mL
  Irinotecan AUC | 3,702 [2,059 to 5,772] | 2,680 [1,626 to 8,492] | 3,957 [3,231 to 4,301] | 2,615 [2,414 to 3,288] | 3,533 [1,906 to 4,301] | 3,121 [2,001 to 7,970]
  APC AUC | 571 [248 to 3,313] | 477 [197 to 1,083] | 511 [293 to 821] | 418 [299 to 457] | 511 [293 to 1,429] | 616 [221 to 985]
  SN-38 AUC | 63.2 [20.5 to 294.6] | 52.9 [28.4 to 119.6] | 80.8 [35.0 to 109.9] | 72.0 [62.6 to 102.0] | 90.0 [35.0 to 235] | 56.7 [26.2 to 398]
  SN-38G AUC | 206.5 [124.3 to 325.3] | 97.6 [53.8 to 243.6] | 141.8 [77.5 to 298.1] | 134.4 [101.1 to 237.8] | 132 [71.0 to 498] | 136 [74.6 to 673]

8. Primary Outcome: Pharmacokinetics When Given Together With Fixed Doses of Irinotecan and Temozolomide in Children and Young Adults With Relapsed or Refractory Neuroblastoma: Irinotecan Clearance
Description: Outcomes included Alisertib, irinotecan, APC, SN-38, and SN-38G. APC, SN-38, and SN-38G are metabolites of irinotecan.
Time Frame: 1st week of cycle 1
Measure: Median (Full Range); unit: L/h
Arm/Group | DL 1 | DL 1B | DL 2B | DL 3B | Ph 2 | Oral Solution
Number analyzed (Participants) | 6 | 6 | 6 | 4 | 12 | 8
L/h | 14.0 [8.8 to 29.4] | 15.7 [4.6 to 27.3] | 10.4 [9.0 to 31.4] | 16.0 [12.6 to 20.1] | 12.6 [7.65 to 31.7] | 10.3 [4.12 to 20.9]

9. Primary Outcome: Response Rate for Patients With Relapsed or Refractory Neuroblastoma Treated With MLN8237, Irinotecan, and Temozolomide at the Identified MTD
Description: Response was graded according to version 1.2 of the NANT response criteria that classifies patients as having one of the following overall response categories based upon underlying response at soft tissue sites, MIBG positive sites, and bone marrow disease: complete response (CR); CR with minimal residual disease (CR-MRD); partial response (PR); minor response (MR); stable disease (SD); and progressive disease (PD). These criteria utilize RECIST criteria for measurable tumors, Curie score for MIBG scan response, and bone marrow (BM) morphology. BM response was graded as CR (required two time points to confirm), CR unconfirmed (one time point only), CR-MRD (bone marrow involvement < 5% at study entry with negative follow-up biopsies), SD, or PD. Patients with at least SD or better underwent central review of MIBG scans, CT scans, and bone marrow pathology slides. Overall responses of CR, CR-MRD, or PR were considered objective responses.
Time Frame: Cycles repeated every 21 days for up to 34 cycles.
Population: The analysis was performed on 19 phase II patients, with 1 inevaluable patient excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Ph 2
Number analyzed (Participants) | 19
Participants
  Complete Response (CR) | 0
  CR-Minimal Residual Disease (MRD) | 0
  Partial Response (PR) | 4
  Minor Response | 2
  Stable Disease | 8
  Progressive Disease | 5
  Response Rate (CR + CR-MRD + PR) | 4

10. Secondary Outcome: Aurora A Expression
Description: To explore whether MYCN status and markers of expression of Aurora A in archival tumor tissue are associated with the antitumor activity of the combination of MLN8237, irinotecan, and temozolomide
Time Frame: From date of study enrollment to the date of progression or withdrawal from the study, up to 34 cycles (about 2 years).
Population: Consisting of patients treated on the Phase 1 (n = 22), Phase 2 (n = 20), and Oral Solution (n = 12) cohorts.
Measure: Number; unit: participants
Groups:
- Objective Responders: Consisting of complete response (CR), CR with minimal residual disease (CR-MRD), and partial response (PR).
- Objective Non-Responders: Consisting of minor response (MR), stable disease (SD) and progressive disease (PD).
Arm/Group | Objective Responders | Objective Non-Responders
Number analyzed (Participants) | 12 | 42
participants
  MYCN Amplified | 1 | 14
  MYCN not Amplified | 9 | 24
  MYCN Missing | 2 | 4
  MYCN Amplified or Myc Positive | 2 | 16
  MYCN Non-amplified and Myc Negative | 5 | 11
  MYCN or Myc Missing | 5 | 15
  Aurora A protein Positive | 2 | 10
  Aurora A protein Negative | 4 | 14
  Aurora A protein Missing | 6 | 18
Statistical Analysis 1: Comparison: Objective Responders vs Objective Non-Responders; Test type: Other; p = 0.14, Fisher Exact — MYCN Amplified vs. MYCN not Amplified
Statistical Analysis 2: Comparison: Objective Responders vs Objective Non-Responders; Test type: Other; p = 0.21, Fisher Exact; MYCN Amplified or Myc Positive vs. MYCN Non-amplified and Myc Negative
Statistical Analysis 3: Comparison: Objective Responders vs Objective Non-Responders; Test type: Other; p = 1.0, Fisher Exact; Aurora A protein Positive vs. Aurora A protein Negative

11. Secondary Outcome: UGT1A1 Genotype
Description: To explore whether UGT1A1 genotype is associated with toxicity in children with refractory neuroblastoma treated with the combination of MLN8237, irinotecan, and temozolomide
Time Frame: Day 7 of cycle 1
Population: Consisting of patients treated on the Phase 1 (n = 22), Phase 2 (n = 20), and Oral Solution (n = 12) cohorts.
Measure: Number; unit: participants
Groups:
- First Cycle DLT Yes: Patients who had DLT in the first cycle of treatment.
- First Cycle DLT No: Patients who did not have DLT in the first cycle of treatment.
- DLT in Any Cycle Yes: Patients who had DLT in any cycle of treatment.
- DLT in Any Cycle No: Patients who did not have DLT in any cycle of treatment.
Arm/Group | First Cycle DLT Yes | First Cycle DLT No | DLT in Any Cycle Yes | DLT in Any Cycle No
Number analyzed (Participants) | 11 | 43 | 27 | 27
participants
  UGT1A1 6\6 | 2 | 15 | 8 | 9
  UGT1A1 6\7 | 3 | 14 | 6 | 11
  UGT1A1 7\7 | 3 | 2 | 4 | 1
  UGT1A1 Missing | 3 | 12 | 9 | 6
Statistical Analysis 1: Comparison: First Cycle DLT Yes vs First Cycle DLT No; Test type: Other; p = 0.094, Fisher Exact — UGT1A1 6\6 vs. UGT1A1 6\7 vs. UGT1A1 7\7
Statistical Analysis 2: Comparison: DLT in Any Cycle Yes vs DLT in Any Cycle No; Test type: Other; p = 0.63, Fisher Exact — UGT1A1 6\6 vs. UGT1A1 6\7 vs. UGT1A1 7\7

12. Secondary Outcome: AURKA Genotype
Description: To explore whether AURKA genotype is associated with antitumor activity in children with refractory neuroblastoma treated with the combination of MLN8237, irinotecan, and temozolomide.
Time Frame: Day 7 of cycle 1
Population: Consisting of patients treated on the Phase 1 (n = 22), Phase 2 (n = 20), and Oral Solution (n = 12) cohorts.
Measure: Number; unit: participants
Arm/Group | Objective Responders | Objective Non-Responders
Number analyzed (Participants) | 12 | 42
participants
  AurkA Codon 31 Summary H | 3 | 9
  AurkA Codon 31 Summary V | 0 | 1
  AurkA Codon 31 Summary W | 5 | 22
  AurkA Codon 31 Summary Missing | 4 | 10
  AurkA Codon 57 Summary H | 3 | 10
  AurkA Codon 57 Summary W | 5 | 22
  AurkA Codon 57 Summary Missing | 4 | 10
Statistical Analysis 1: Comparison: Objective Responders vs Objective Non-Responders; Test type: Other; p = 0.90, Fisher Exact — AurkA Codon 31 Summary H vs. AurkA Codon 31 Summary V vs. AurkA Codon 31 Summary W
Statistical Analysis 2: Comparison: Objective Responders vs Objective Non-Responders; Test type: Other; p = 1.0, Fisher Exact — AurkA Codon 57 Summary H vs. AurkA Codon 57 Summary W

13. Secondary Outcome: One Year Progression Free Survival Rate
Description: To determine the progression free survival rates for patients with relapsed or refractory neuroblastoma treated with MLN8237, irinotecan, and temozolomide at the identified MTD
Time Frame: 1 Years after completion of study
Population: The analysis was performed in phase II patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Ph 2
Number analyzed (Participants) | 20
Participants | 4

ADVERSE EVENTS:
Time Frame: From date of study enrollment to the date of progression or withdrawal from the study, up to 34 cycles (about 2 years).
Arm/Group | DL 1 | DL 1B | DL 2B | DL 3B | Ph 2 | Oral Solution
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/4 | 0/20 | 0/12
Serious Adverse Events (participants affected / at risk) | 3/6 | 3/6 | 3/6 | 2/4 | 1/20 | 2/12
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 4/4 | 20/20 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DL 1 (N=6) | DL 1B (N=6) | DL 2B (N=6) | DL 3B (N=4) | Ph 2 (N=20) | Oral Solution (N=12)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Movements involuntary (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DL 1 (N=6) | DL 1B (N=6) | DL 2B (N=6) | DL 3B (N=4) | Ph 2 (N=20) | Oral Solution (N=12)
Anemia (Blood and lymphatic system disorders) | 6 (50) | 6 (61) | 6 (100) | 4 (17) | 19 (147) | 10 (41) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (4) | 2 (2) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Palpitations (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 6 (22) | 1 (3) | 4 (9) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Ear pain (Ear and labyrinth disorders) | 2 (5) | 0 (0) | 2 (2) | 1 (5) | 0 (0) | 1 (1) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (14) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Blurred vision (Eye disorders) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 2 (13) | 1 (1) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 2 (3) | 1 (1) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Abdominal pain (Gastrointestinal disorders) | 4 (17) | 2 (8) | 5 (20) | 0 (0) | 10 (17) | 4 (9) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Anal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (5) | 1 (2) | 0 (0) | 2 (2) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Diarrhea (Gastrointestinal disorders) | 6 (45) | 6 (27) | 6 (50) | 4 (14) | 18 (88) | 9 (27) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 3 (5) | 2 (2) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Mucositis oral (Gastrointestinal disorders) | 2 (3) | 1 (1) | 4 (18) | 2 (2) | 5 (11) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Nausea (Gastrointestinal disorders) | 6 (33) | 5 (37) | 5 (52) | 4 (11) | 18 (98) | 9 (17) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Rectal hemorrhage (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (5) | 1 (1) | 1 (2) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (3) | 1 (4) | 0 (0) | 1 (2) | 1 (1) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Vomiting (Gastrointestinal disorders) | 4 (29) | 6 (38) | 6 (34) | 4 (6) | 17 (68) | 11 (24) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Chills (General disorders) | 1 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Edema face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Edema trunk (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Fatigue (General disorders) | 4 (10) | 3 (6) | 5 (24) | 3 (12) | 10 (23) | 4 (7) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Fever (General disorders) | 5 (7) | 3 (10) | 5 (9) | 2 (2) | 10 (15) | 4 (4) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Irritability (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 3 (4) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain (General disorders) | 2 (3) | 1 (1) | 1 (5) | 1 (1) | 3 (6) | 2 (3) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Conjunctivitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 1 (2) | 2 (6) | 1 (1) | 3 (3) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Otitis externa (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Rhinitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Upper respiratory infection (Infections and infestations) | 0 (0) | 2 (4) | 3 (8) | 1 (1) | 6 (8) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (4) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 3 (7) | 1 (2) | 4 (9) | 1 (3) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Alanine aminotransferase increased (Investigations) | 6 (36) | 4 (32) | 5 (51) | 3 (3) | 18 (112) | 8 (23) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Alkaline phosphatase increased (Investigations) | 2 (4) | 0 (0) | 1 (6) | 0 (0) | 7 (32) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Aspartate aminotransferase increased (Investigations) | 6 (42) | 4 (23) | 6 (51) | 2 (2) | 17 (103) | 10 (22) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Blood bilirubin increased (Investigations) | 2 (17) | 2 (11) | 1 (7) | 1 (2) | 3 (4) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Creatinine increased (Investigations) | 0 (0) | 2 (5) | 3 (27) | 1 (1) | 5 (9) | 3 (4) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
GGT increased (Investigations) | 3 (12) | 1 (32) | 2 (3) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hemoglobin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Investigations - Other, specify (Investigations) | 0 (0) | 0 (0) | 1 (5) | 1 (2) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Lymphocyte count decreased (Investigations) | 3 (32) | 4 (21) | 5 (43) | 3 (14) | 17 (111) | 10 (26) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Lymphocyte count increased (Investigations) | 1 (2) | 0 (0) | 2 (8) | 0 (0) | 1 (2) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Neutrophil count decreased (Investigations) | 6 (43) | 6 (46) | 6 (66) | 4 (15) | 20 (132) | 12 (41) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Platelet count decreased (Investigations) | 5 (43) | 5 (55) | 6 (93) | 4 (16) | 20 (154) | 10 (43) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Weight gain (Investigations) | 0 (0) | 0 (0) | 2 (25) | 0 (0) | 1 (3) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Weight loss (Investigations) | 2 (22) | 1 (1) | 2 (13) | 3 (4) | 3 (9) | 5 (6) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
White blood cell decreased (Investigations) | 6 (55) | 6 (57) | 6 (89) | 3 (15) | 20 (150) | 11 (45) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 1 (1) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Anorexia (Metabolism and nutrition disorders) | 3 (7) | 2 (3) | 4 (40) | 4 (9) | 10 (25) | 5 (17) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 1 (4) | 4 (6) | 1 (1) | 6 (10) | 2 (4) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hyperglycemia (Metabolism and nutrition disorders) | 4 (11) | 2 (5) | 4 (22) | 2 (3) | 9 (27) | 5 (9) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hyperkalemia (Metabolism and nutrition disorders) | 1 (4) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (17) | 0 (0) | 0 (0) | 3 (11) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (10) | 0 (0) | 3 (6) | 3 (4) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (18) | 3 (5) | 5 (18) | 2 (2) | 11 (19) | 8 (14) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hypocalcemia (Metabolism and nutrition disorders) | 3 (27) | 1 (2) | 5 (29) | 1 (1) | 11 (22) | 5 (9) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hypoglycemia (Metabolism and nutrition disorders) | 2 (3) | 3 (13) | 2 (2) | 0 (0) | 1 (4) | 1 (1) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hypokalemia (Metabolism and nutrition disorders) | 4 (29) | 3 (6) | 4 (14) | 3 (4) | 10 (26) | 6 (7) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2) | 2 (9) | 2 (10) | 2 (2) | 5 (10) | 4 (4) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hyponatremia (Metabolism and nutrition disorders) | 4 (11) | 2 (10) | 5 (9) | 2 (3) | 8 (12) | 6 (6) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (7) | 1 (2) | 2 (5) | 1 (1) | 8 (11) | 6 (15) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 1 (2) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (3) | 4 (25) | 1 (2) | 4 (5) | 3 (4) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (9) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Depressed level of consciousness (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 4 (4) | 2 (2) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Headache (Nervous system disorders) | 2 (3) | 3 (9) | 3 (11) | 3 (6) | 9 (18) | 1 (1) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Somnolence (Nervous system disorders) | 1 (7) | 2 (3) | 0 (0) | 2 (2) | 4 (4) | 3 (4) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Agitation (Psychiatric disorders) | 1 (3) | 1 (8) | 0 (0) | 2 (3) | 2 (2) | 2 (3) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Anxiety (Psychiatric disorders) | 0 (0) | 2 (9) | 2 (5) | 1 (2) | 3 (9) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 3 (24) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (23) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Urine discoloration (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Penile pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (8) | 0 (0) | 2 (6) | 1 (8) | 3 (13) | 1 (14) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (10) | 5 (13) | 5 (29) | 3 (9) | 7 (14) | 5 (9) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (6) | 5 (16) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 3 (5) | 3 (10) | 1 (2) | 6 (7) | 1 (3) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (22) | 1 (2) | 2 (2) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 2 (5) | 1 (2) | 4 (7) | 1 (2) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Alopecia (Skin and subcutaneous tissue disorders) | 3 (38) | 1 (2) | 3 (52) | 2 (12) | 8 (86) | 4 (32) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Dry skin (Skin and subcutaneous tissue disorders) | 1 (5) | 0 (0) | 3 (9) | 0 (0) | 2 (8) | 1 (18) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Pruritus (Skin and subcutaneous tissue disorders) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (4) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (3) | 2 (7) | 1 (1) | 3 (3) | 2 (3) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (11) | 0 (0) | 1 (2) | 2 (2) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (12) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (4) | 0 (0) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (7) | 1 (2) | 2 (7) | 1 (1) — As requested, we are reporting all toxicities of all grades, whether or not they are related to the regimen or known to be related to non-treatment causes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/35/NCT01601535/Prot_SAP_ICF_000.pdf